CLINICAL TRIAL: NCT07213297
Title: Comprehensive Program for Hereditary Transthyretin Amyloidosis
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital de Alta Complejidad en Red (Other)
Responsible Party: Principal Investigator, Gisela Mariel Zanga, PRINCIPAL INVESTIGATOR, Hospital de Alta Complejidad en Red
Other Study IDs: ESCAN
Record Dates: First submitted 2025-09-05; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Amyloidosis in Transthyretin (TTR); Amyloidosis, Familial
Keywords: transthyretin; amyloidosis; comprensive care
MeSH Terms: conditions — Amyloidosis, Familial; Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants over 18 years of age diagnosed with hereditary transthyretin amyloidosis: Participants with a pathogenic variant of the TTR gene confirmed by genetic testing, whether symptomatic and/or with suspected disease progression, as well as asymptomatic carriers of these variants, will be included. Individuals with wild-type TTR amyloidosis will be excluded .
  Interventions: Other: clinical assessments and complementary examinations

INTERVENTIONS:
Other: clinical assessments and complementary examinations — Evaluation Plan
  Comprehensive Examination: Complete medical history and physical examination of all body systems, including height and weight measurements.
  Clinical Parameters: Pulse/heart rate, respiratory rate, and SpO2 will be monitored. The NYHA classification will be used to assess heart failure if applicable.
  Neurological Examination: Includes motor strength testing, sensory testing (pinprick, light touch, temperature, proprioception), deep tendon reflexes, and gait assessment.
  Electrocardiogram (ECG): A 12-lead ECG will be performed with the subject at rest for at least 5 minutes in a supine position.
  24-hour Holter Monitoring: Conducted in cases of suspected arrhythmias or echocardiographic findings indicating arrhythmias.
  Color Dosments and complementary examinations

SUMMARY:
The Comprehensive Program for Hereditary Transthyretin Amyloidosis describes a prospective observational study focused on understanding hereditary transthyretin amyloidosis (ATTR), a progressive and potentially fatal condition marked by amyloid fibril deposits impacting multiple organs. The trial aims to characterize patient phenotypes, investigate factors affecting disease progression, and identify minimum criteria for disease onset. Conducted at Néstor Kirchner Hospital, the trial enrolls participants over 18 years old with confirmed pathogenic TTR variants. It includes thorough evaluations such as genetic testing sponsored by pharmaceutical companies, clinical assessments, and diverse diagnostic tests.

ELIGIBILITY:
Inclusion Criteria:

-Participants with a pathogenic variant of the TTR gene (Hereditary Amyloidosis)

Exclusion Criteria:

* wild-type TTR amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants over 18 years of age diagnosed with hereditary transthyretin amyloidosis with a pathogenic variant of the TTR gene confirmed by genetic testing, whether symptomatic and/or with suspected disease progression, as well as asymptomatic carriers of these variants, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Phenotypic classification | 3 YEARS
  1. Predominantly Cardiac Phenotype: Patients will present with abnormal electrocardiograms (ECG) due to rhythm disturbances, heart failure, or dyspnea.
     They will exhibit no more than mild neurological or gastrointestinal (GI) symptoms.
     Conditions such as erectile dysfunction, constipation, and carpal tunnel syndrome will be excluded from this phenotype.
  2. Predominantly Neurological Phenotype: Patients will exhibit neurological or GI symptoms of any severity. They will not have abnormal ECGs due to rhythm disturbances, heart failure, or dyspnea.
  Neurological and GI symptoms will need to be continuous and definitively linked to amyloidosis.
  3]) Mixed Phenotype: Patients will present with abnormal ECGs due to rhythm disturbances, heart failure, or dyspnea.
  They will also have neurological or GI symptoms of any severity. These patients will not meet the criteria for a predominantly cardiac or neurological phenotype.

SECONDARY OUTCOMES:
Change from baseline in New York Heart Association (NYHA) functional class | 3 years
  Functional class assessed using the NYHA scale (range I-IV, higher class indicates worse cardiac function).
Change from baseline in 6-Minute Walk Test (6MWT) distance | 3 years
  Distance walked in meters will be measured according to ATS guidelines. Lower values indicate reduced functional capacity
Change from baseline in N-terminal pro-brain natriuretic peptide (Pro-BNP) | 3 years
  Serum concentration measured in pg/mL. Higher values indicate worse cardiac function.
Change from baseline in Troponin T | 3 years
  Serum concentration measured in ng/L. Higher values indicate myocardial injury
Change from baseline in Microalbuminuria | 3 years
  Urinary albumin excretion measured in mg/24h. Higher values indicate worse renal involvement.
Change from baseline in Left Ventricular Ejection Fraction | 3 years
  Ejection fraction (%) measured by echocardiography. Lower values indicate worse cardiac function
Change from baseline in Left Ventricular Wall Thickness | 3 years
  Wall thickness measured in millimeters by echocardiography. Higher values indicate worse disease progression.
Change from baseline in diastolic dysfunction grade | 3 years
  Diastolic dysfunction assessed by echocardiography following ASE guidelines. Higher grade indicates worse dysfunction.
Incidence of atrial fibrillation, atrioventricular block, or PR interval prolongation | 3 years
  Presence of atrial fibrillation, new AV block, or PR interval prolongation assessed by ECG. Categorical outcome (Yes/No).
Change from baseline in Coutinho/PND (Polyneuropathy Disability) score | 3 years
  Score range 0-IV; higher score indicates greater disability
Change from baseline in Neuropathy Impairment Score (NIS) | 3 years
  Total score range 0-244; higher values indicate worse neuropathy.
Change from baseline in COMPASS-31 total score | 3 years
  Questionnaire score range 0-100; higher values indicate worse autonomic symptoms.
Change from baseline in Norfolk QoL-DN score | 3 years
  Total score range -4 to 136; higher values indicate worse quality of life related to neuropathy.
Change from baseline in RODS (Rasch-built Overall Disability Scale) | 3 years
  Score range 0-48; lower values indicate greater disability
Change from baseline in Body Mass Index (BMI) | 3 years
  BMI calculated as weight (kg)/height (m²). Both weight and height will be measured and aggregated to report BMI. Higher or lower values may reflect disease progression.

OTHER OUTCOMES:
Minimum criteria | 3 years
  To explore minimum criteria for disease onset in patients initially considered asymptomatic:
  1. A quantified symptom or sign definitely related to the onset of the disease.
     * Sensorimotor neuropathy
     * Autonomic neuropathy
     * Heart involvement
     * Kidney or eye involvement either
  2. Any likely related symptoms plus 1 abnormal test result. either
  3. Absence of symptoms and 2 abnormal test results

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Cuenca Alta de Cañuelas, Cañuelas, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pinto MV, Barreira AA, Bulle AS, Freitas MRG, Franca MC Jr, Gondim FAA, Marrone CD, Marques W Jr, Nascimento OJM, Rotta FT, Pupe C, Waddington-Cruz M. Brazilian consensus for diagnosis, management and treatment of transthyretin familial amyloid polyneuropathy. Arq Neuropsiquiatr. 2018 Sep;76(9):609-621. doi: 10.1590/0004-282X20180094. PMID 30365625